CLINICAL TRIAL: NCT05970718
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses of REGN7544, an Antagonistic Monoclonal Antibody to NPR1, in Healthy Adults
Brief Title: A Trial to Learn if Different Doses of REGN7544 Are Safe in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R7544-HV-22109
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Healthy Volunteers
Keywords: Hypotension and/or hypovolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- IV Dose Level 1 (Experimental): Randomized 6:2 for single ascending IV dose
  Interventions: Drug: REGN7544; Drug: Matching Placebo
- IV Dose Level 2 (Experimental): Randomized 6:2 for single ascending IV dose
  Interventions: Drug: REGN7544; Drug: Matching Placebo
- IV Dose Level 3 (Experimental): Randomized 6:2 for single ascending IV dose
  Interventions: Drug: REGN7544; Drug: Matching Placebo
- IV Dose Level 4 (Experimental): Randomized 6:2 for single ascending IV dose
  Interventions: Drug: REGN7544; Drug: Matching Placebo
- IV Dose Level 5 (Experimental): Randomized 6:2 for single ascending IV dose
  Interventions: Drug: REGN7544; Drug: Matching Placebo
- IV Dose Level 6 (Experimental): Randomized 6:2 for single ascending IV dose
  Interventions: Drug: REGN7544; Drug: Matching Placebo
- SC Dose Level 1 (Experimental): Randomized 6:2 for single ascending SC dose
  Interventions: Drug: REGN7544; Drug: Matching Placebo
- SC Dose Level 2 (Experimental): Randomized 6:2 for single ascending SC dose
  Interventions: Drug: REGN7544; Drug: Matching Placebo
- SC Dose Level 3 (Experimental): Randomized 6:2 for single ascending SC dose
  Interventions: Drug: REGN7544; Drug: Matching Placebo
- Optional Cohort 1 (Experimental): Randomized 6:2 for single ascending dose This is an optional cohort, that may be IV or SC and will not exceed highest dose level
  Interventions: Drug: REGN7544; Drug: Matching Placebo
- Optional Cohort 2 (Experimental): Randomized 6:2 Randomized 6:2 for single ascending dose This is an optional cohort, that may be IV o SC and will not exceed highest dose level
  Interventions: Drug: REGN7544; Drug: Matching Placebo

INTERVENTIONS:
Drug: REGN7544 — Solution for single ascending Intravenous (IV) or Subcutaneous (SC) administration
Drug: Matching Placebo — Solution for single ascending IV or SC administration per the protocol

SUMMARY:
The study is researching an experimental drug called REGN7544.The study is focused on healthy adults. The aim of the study is to see how safe and tolerable the study drug is in healthy adults.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in your blood at different times
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Has a body mass index between 18 and 32 kg/m^2
2. Is judged by the investigator to be in good health based on medical history, physical examination, vital sign measurements, and electrocardiograms (ECGs) performed at screening and/or prior to administration of initial dose of study drug, as defined in the protocol
3. Has normal blood pressure (BP) and pulse rate readings, as defined in the protocol
4. Difference between semi-recumbent systolic blood pressure (SBP) measurements in left and right arm less than 20 mmHg at screening visit

Key Exclusion Criteria:

1. History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric or neurological disease, as assessed by the investigator that may confound the results of the study or poses an additional risk to the participant by study participation
2. History, in the past 2 years of a diagnosis of hypertension, symptomatic hypotension (BP <90/50 mmHg with associated symptoms), symptomatic orthostatic hypotension, postural orthostatic tachycardia syndrome, syncope, or clinically significant cardiac arrhythmia
3. Presents any concern to the study investigator that might confound the results of the study or poses an additional risk to the participant by their participation in the study
4. Was hospitalized (ie, >24 hours) for any reason within 30 days of screening
5. Is a current smoker or former smoker, including e-cigarettes, who stopped smoking within 3 months prior to screening

NOTE: Other protocol defined inclusion / exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) | Through approximately day 162
Severity of TEAEs | Through approximately day 162

SECONDARY OUTCOMES:
Changes from baseline in Systolic Blood Pressure (SBP) | Through day 6
Changes from baseline in Diastolic Blood Pressure (DBP) | Through day 6
Changes from baseline in Mean Arterial Pressure (MAP) | Through day 6
Changes from baseline in Pulse Pressure (PP) | Through day 6
Concentrations of REGN7544 in serum over time | Through approximately day 162
Incidence of treatment-emergent Anti-Drug Antibody (ADA) | Through approximately day 162
Titer of ADA | Through approximately day 162

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- New Zealand Clinical Research, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/